CLINICAL TRIAL: NCT00552968
Title: Pain Prevalence in the Trauma Population at Sunnybrook Hospital
Brief Title: Pain Prevalence in the Trauma Population
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Lynn Haslam, Nurse Practitioner, Dept of Anesthesia, Sunnybrook Health Sciences Centre
Other Study IDs: 208-2007
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Trauma
Keywords: trauma; pain
MeSH Terms: conditions — Wounds and Injuries; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The incidence of pain in the post traumatic population is an area that has little to no investigation. This study seeks to determine the incidence and experience of pain in this vulnerable population at different time points - while in hospital, 4 weeks post injury, 3 months post injury.

DETAILED DESCRIPTION:
This pilot study will be a convenience sample from trauma inpatients at the Sunnybrook Campus. The purpose of the study is twofold: to investigate the prevalence of chronic pain that develops in the trauma population at Sunnybrook, and to see if neuropathic pain exists in this population, acute and/or chronically.

ELIGIBILITY:
Inclusion Criteria:

* Over 16 years of age
* ability to read / write in English
* ability to complete an informed consent

Exclusion Criteria:

* history of chronic pain
* unable to give informed consent
* unable to read / write English

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have been admitted to hospital due to a traumatic injury.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of pain at 3 months post traumatic injury. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Haslam, RN MN ACNP, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada